CLINICAL TRIAL: NCT06010264
Title: THE EFFECTS OF EARLY PERIOD KINESIO TAPE ON CLINICAL OUTCOMES IN PATIENTS WITH ARTROSCOPIC ROTATOR CUFF REPAIR
Brief Title: THE EFFECTS OF EARLY PERIOD KINESIOTAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Muhammed İhsan KODAK, PHD / LECTURER, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14/123
Record Dates: First submitted 2023-08-10; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Rotator Cuff Injuries; Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesiotaping group (Experimental): Kinesiotaping + Standard Physiotherapy Program
  Interventions: Other: Kinesiotape
- Control group (Active Comparator): Standard Physiotherapy Program
  Interventions: Other: Standard Physiotherapy Program
- Shamtape Group (Sham Comparator): Shamtaping + Standard Physiotherapy Program
  Interventions: Other: Shamtape

INTERVENTIONS:
Other: Kinesiotape — In the kinesiotaping group, kinesiotape was applied from the first postoperative day in addition to conservative treatment.
  Kinesiobant application was performed regularly until the 6th week by a researcher with a certificate in kinesiobanting in accordance with the lymphatic correction and pain inhibition techniques described by Kenzo Kase.
  Conservative Treatment Program. 1-10 days: Patient education Pendulum exercises Active hand and wrist exercises Cold Application 1-6 Weeks: Pendulum exercises are continued Active hand and wrist exercises are continued Cold application is continued Passive arm elevation with opposite hand support in supine position Elbow flexion/extension exercise at the limit of pain
  Arms: Kinesiotaping group
Other: Shamtape — In the sham taping group, sham tape was applied from the first postoperative day in addition to conservative treatment. Medical flasters were used as sham tape. Sham tapes were applied by cutting in the same fan shape as in kinesioband.
  Conservative Treatment Program. 1-10 days: Patient education Pendulum exercises Active hand and wrist exercises Cold Application 1-6 Weeks: Pendulum exercises are continued Active hand and wrist exercises are continued Cold application is continued Passive arm elevation with opposite hand support in supine position Elbow flexion/extension exercise at the limit of pain
  Arms: Shamtape Group
Other: Standard Physiotherapy Program — Conservative Treatment Program. 1-10 days: Patient education Pendulum exercises Active hand and wrist exercises Cold Application 1-6 Weeks: Pendulum exercises are continued Active hand and wrist exercises are continued Cold application is continued Passive arm elevation with opposite hand support in supine position Elbow flexion/extension exercise at the limit of pain
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to the effects of kinesio tape application on pain, edema, range of motion and functionality .

The main questions it aims to answer are:

* Does kinesiotape application reduce pain and edema and improve quality of life in the early period in individuals undergoing arthroscopic rotator cuff repair?
* Does kinesiotape application provide early restoration of functional activity level in individuals undergoing arthroscopic rotator cuff repair?

Participants will receive kinesiotaping in addition to traditional physiotherapy programs.

If there is a comparison group: Researchers will compare kinesiotape group, shamtape group and control group to see if kinesiotaping.

DETAILED DESCRIPTION:
Chronic shoulder pain is the second most common musculoskeletal problem in the population with a prevalence ranging from 15% to 22%. Rotator cuff (RM) tears are one of the important pathophysiologic conditions leading to shoulder pain. Early treatment of RM tears is conservative and includes oral analgesics, non-steroidal anti-inflammatory drugs, corticosteroid injections if necessary and physiotherapy methods. Treatment of rotator sheath problems may be surgical and/or conservative depending on the indications. Surgical treatment is inevitable for partial tears and complete ruptures that do not respond to conservative treatment. After surgery, a good rehabilitation program is needed to increase the success of the surgical intervention, return to functional activities and improve the patient's quality of life. One of the most important problems for the patient, physician and physiotherapist in the rehabilitation program to be applied in this period is the immobilization period of 6 weeks. This is the recommended time for tissue healing. However, the negative effects of prolonged immobilization should not be forgotten. It is important to use early physiotherapy applications to prevent adhesions and reduce complications that may occur.

The Kinesio Taping® technique and Kinesio Tex® tape were developed in 1973 by Dr. Kenzo Kase, a Japanese chiropractor and acupuncturist. There is an increasing number of health professionals, including physicians and physiotherapists who deal with musculoskeletal diseases and lymphology, who apply this method to their patients all over the world. It is also widely used in the sports world, especially considering its ease of use and effects. It helps structures such as the musculoskeletal system, circulatory system and nervous system to return to normal function. It is a preferred method because these bands are easy to apply and patients can easily remove them. In the literature, there is no study examining the effects of kinesio tape application after rotator cuff repair.

Considering the effects of kinesio tape on pain and edema; we think that it will have positive results in the rehabilitation program applied after rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65,
* Arthroscopic rotator cuff repair as a surgical method,
* diagnosis of a small or medium-sized (<3 cm) rotator cuff tear by magnetic resonance imaging,
* Having a score above 24 on the Mini Mental State Examination,
* Volunteering to participate in the study.

Exclusion Criteria:

* Presence of diabetes mellitus,
* Stage three and above according to the Goutallier fatty degeneration classification,
* Presence of a neurological problem,
* Presence of cervical disc herniation,
* Past history of orthopedic disease on the affected side,
* Presence of osteoarthritis, rheumatoid arthritis or other systemic inflammatory problem,
* Corticosteroid injection for the affected side within 6 weeks before diagnosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Pain severity | 7 weeks
  Visual Analogue Scale (0-10, higher means worse)
Edema | 7 weeks
  Diameter measurement was performed to evaluate the level of edema in the shoulder joint. Two reference points, the posterosuperior end of the acromion and the korkoid process, were used to measure the diameter of the shoulder. First, the distance between these points on the upper border of the deltoid muscle was measured with a tape measure and recorded. The second measurement was taken 1 cm lateral to the first measurement, over the middle deltoid and recorded.

SECONDARY OUTCOMES:
Modified Constant-Murley score | 7 weeks
  The Modified Constant-Murley score is a 100-point scoring system that is divided into 4 subscales: pain, 15 points; activities of daily living (ADL), 20; range of motion (ROM), 40; and strength, 25. The pain and ADL subscales are self-reported by the patient. In the original version, the pain score was graded as none = 15, mild = 10, moderate = 5, and severe = 0.
REVISED OXFORD SHOULDER SCORE | 7 weeks
  REVISED OXFORD SHOULDER SCORE was developed to evaluate the functional parameters of the shoulder after surgery. It consists of a total of 12 questions. Each question has 5 answers ranging from 0 (bad score) to 4 (good score). The total score ranges from 0 to 48. 0 indicates the worst result, while the higher the score, the better the functionality. A score between 0-19 indicates severe disability, 20-29 indicates moderate disability, 30-39 indicates mild disability. A score between 40-48 indicates adequate functionality.
SHOULDER PAIN AND DISABILITY INDEX | 7 weeks
  The SPADI is a 13 item self-reported questionnaire assessing pain and functional status. Each item is measured on a 0-10 scale and a 0-100 score calculated. Higher scores represent greater levels of pain and disability. The SPADI has been shown to have good test-re-test reliability and be sensitive to change.
Western Ontario Rotator Cuff Index | 7 weeks
  WORC consists of 5 sections with 21 questions. The answer to each question is given on the VAS. The final score is between 0 and 2100. The higher the score, the lower the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırsehir Ahi Evran Universty, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reynard F, Vuistiner P, Leger B, Konzelmann M. Immediate and short-term effects of kinesiotaping on muscular activity, mobility, strength and pain after rotator cuff surgery: a crossover clinical trial. BMC Musculoskelet Disord. 2018 Aug 22;19(1):305. doi: 10.1186/s12891-018-2169-5. PMID 30134883
- [Result] Gulenc B, Yalcin S, Genc SG, Bicer H, Erdil M. Is Kinesiotherapy Effective in Relieving Pain and Reducing Swelling after Shoulder Arthroscopy? Acta Chir Orthop Traumatol Cech. 2019;86(3):216-219. PMID 31333187